CLINICAL TRIAL: NCT02512809
Title: Isoflurane-induced Neuroinflammation in Children With Hydrocephalus: A Bench-to-bedside, Translational Study of Molecular Pathways and Therapeutic Approaches
Brief Title: Isoflurane-induced Neuroinflammation in Children With Hydrocephalus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI moving to another institution.
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB14-00625
Record Dates: First submitted 2015-02-23; First posted 2015-07-31 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Toxicity; Hydrocephalus
MeSH Terms: conditions — Hydrocephalus | interventions — Isoflurane; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isoflurane Arm (Experimental): Pediatric patients, aged 0-5 years, diagnosed with hydrocephalus undergoing a surgical (non-bedside) shunting procedure with general anesthesia. Pts will receive a standardized general anesthetic with isoflurane.
  Interventions: Drug: Isoflurane
- Dexmedetomidine/remifentanil Arm (Experimental): Pediatric patients, aged 0-5 years, diagnosed with hydrocephalus undergoing a surgical (non-bedside) shunting procedure with general anesthesia. Pts will receive a standardized general anesthetic with dexmedetomidine and remifentanil infusions..
  Interventions: Drug: Dexmedetomidine
- MRI Control Arm (No Intervention): Otherwise healthy pediatric patients, aged 0-5 years, undergoing MRI with general anesthesia for evaluation of non-neurologic disease. Patients will receive a standardized general anesthetic with isoflurane.

INTERVENTIONS:
Drug: Isoflurane
  Other Names: Isosthesia, Forane
  Arms: Isoflurane Arm
Drug: Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine/remifentanil Arm

SUMMARY:
The investigators will quantify inflammatory biomarkers in cerebrospinal fluid (CSF) and serum of children with hydrocephalus who are undergoing ventriculoperitoneal shunt placement under isoflurane anesthesia.

DETAILED DESCRIPTION:
Background & Significance. Each year, millions of children receive general anesthesia. Isoflurane, a GABA type A (GABAA) receptor agonist is an inhaled anesthetic commonly used in clinical anesthesia practice worldwide. Anesthetics traditionally have been assumed to be safe as long as severe hypotension and hypoxia are avoided. Interfering with the balance of excitatory and inhibitory neurotransmitters in the developing brain may interfere with the formation of synaptic connections and enhance the normal apoptotic processes that lead to neuronal pruning and may induce neuroinflammation. Such enhanced neuronal pruning and neuroinflammation could lead to excessive neuronal loss at critical times during brain development and consequently cause later learning disabilities. Recent reports of neurotoxicity induced with isoflurane have triggered significant concern about the safety of this agent.

Investigations into neuroinflammation and apoptosis after anesthetic exposure in human children have been limited due to ethical and methodological concerns. Studies that have been done have been largely retrospective, population-based studies. Results from these studies have been mixed, some showing a decline in neurocognitive performance, some showing no change. Further, the vast majority of prospective, hypothesis-driven research has been undertaken in animal models. Developing a clinically relevant animal model and testing resultant hypotheses in humans are critical steps in determining the underlying cause of these changes as well as identifying possible therapeutic targets. The investigators hypothesize that piglets exposed to commonly used anesthetics will exhibit increased neuroinflammation when compared with controls. It is further hypothesized children undergoing neurosurgery with isoflurane anesthesia will show evidence of increased central nervous system inflammation. Finally, the investigators hypothesize that significantly less robust inflammation will be seen in patients undergoing MRI with general anesthesia (no surgery), indicating a role of surgical stress in the modulation of isoflurane-induced neuroinflammation.

Clinical/Translational Investigation (NCH): Surgery Group. Patients aged 0-5 years undergoing general anesthesia for ventriculoperitoneal shunt (VPS) repair will have CSF and serum sampled at the beginning of surgery (after induction but before surgical incision) and at the end of surgery (after closure but before emergence). Each of these patients will be randomized to a standardized anesthetic. An additional CSF sample will be taken prior to post anesthesia care unit (PACU) discharge. These samples will be analyzed as described above. Control Group. Patients undergoing diagnostic MRI under general anesthesia for non-neurologic pathology will receive a standardized anesthetic. Serum will be collected at the beginning and end of the procedure and will be analyzed for inflammation as above.

Short term goals: Demonstrate that isoflurane has a role in modulation of neuroinflammation in humans. Determine if surgical stress also has a role in modulation of this inflammation. Develop a clinically relevant animal model for hypothesis-driven anesthetic neuroinflammation research.

Long term goals: Identify which anesthetic regimens, if any, are safe for use in the developing brain. Identify therapeutic targets for prevention or treatment of anesthetic-induced neuroinflammation. Obtain independent federal funding for future research and establish an experimental neuroscience program on the Nationwide Children's campus.

ELIGIBILITY:
Inclusion Criteria (HC study patients):

* Pediatric patients, aged 6 months-less than 11 years, diagnosed with hydrocephalus undergoing a primary surgical (non-bedside) shunting procedure with general anesthesia.
* Participants must have a parent/guardian who is able to provide written informed consent in accordance with human investigation committee guidelines.
* The shunting procedure must be an initial VPS placement (not a VPS revision).

Inclusion Criteria (MRI with general anesthesia: peripheral blood patients; anesthesia but no surgery):

* Otherwise healthy pediatric patients, aged 6 months-less than 11 years, undergoing MRI with general anesthesia for evaluation of non-neurologic, non-inflammatory disease.
* Participants must have a parent/guardian who is able to provide written informed consent in accordance with IRB guidelines.

Exclusion Criteria (HC study patients):

* Any active infection or infection within the last 14 days.
* Treatment in the last 48 hours with non-steroidal anti-inflammatory (NSAID) or corticosteroid medications.
* Anticoagulant administration in the last 48 hours.
* Treatment with any drug known to induce or suppress inflammation.
* Clinically unstable patients.
* Patients that have an American Society of Anesthesiologists physical status ≥4 (severe, life-threatening disease).
* Infants born more than 4 weeks premature.

Exclusion Criteria (MRI with general anesthesia: peripheral blood patients; anesthesia but no surgery):

* Known central nervous system disease.
* Treatment in the last 48 hours with non-steroidal anti-inflammatory (NSAID) or corticosteroid medications.
* Treatment with any drug known to induce or suppress inflammation.
* Patients that have an American Society of Anesthesiologists (ASA) physical status ≥4 (severe, life-threatening disease).
* Infants born more than 4 weeks premature.

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tobias, M.D., Principal Investigator — Nationwide Children's Hospital

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no participants assigned to the "Isoflurane" and "Dexmedetomidine/Remifentanil Arm" Arms/Groups as only the MRI control arm completed enrollment prior to the original PI leaving the institution and there was no enrollment in the other 2 arms.
Period: Overall Study
Arm/Group | MRI Control Arm
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only the MRI control arm completed enrollment prior to the original PI leaving the institution. There was no enrollment in the other 2 arms.
Groups:
- Isoflurane Arm: Pediatric patients, aged 0-5 years, diagnosed with hydrocephalus undergoing a surgical (non-bedside) shunting procedure with general anesthesia. Pts will receive a standardized general anesthetic with isoflurane.
  Isoflurane
- Dexmedetomidine/Remifentanil Arm: Pediatric patients, aged 0-5 years, diagnosed with hydrocephalus undergoing a surgical (non-bedside) shunting procedure with general anesthesia. Pts will receive a standardized general anesthetic with dexmedetomidine and remifentanil infusions..
  Dexmedetomidine
- Total: Total of all reporting groups
Arm/Group | Isoflurane Arm | Dexmedetomidine/Remifentanil Arm | MRI Control Arm | Total
Number analyzed (Participants) | 0 | 0 | 25 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 25 | 25
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 3.73 (2.49) | 3.73 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 10 | 10
  Male |  |  | 15 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0
  Asian |  |  | 3 | 3
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
  Black or African American |  |  | 1 | 1
  White |  |  | 21 | 21
  More than one race |  |  | 0 | 0
  Unknown or Not Reported |  |  | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] |  |  | 17.4 (8.3) | 17.4 (8.3)
Anesthetic Time [Mean (Standard Deviation); unit: minutes] |  |  | 54.7 (24.7) | 54.7 (24.7)
Previous Anesthesia [Count of Participants; unit: Participants]
  Yes |  |  | 12 | 12
  No |  |  | 13 | 13
American Society of Anesthesiologists (ASA) Physical Status classification [Count of Participants; unit: Participants] — ASA 1: Normal healthy patient
  ASA 2: Patients with mild systemic disease
  ASA 3: Patients with severe systemic disease
  ASA 4: Patients with severe systemic disease that is a constant threat to life
  ASA 5: Moribund patients who are not expected to survive without the operation
  ASA 6: A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA 1 |  |  | 8 | 8
    ASA 2 |  |  | 17 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Cytokine Levels
Description: Surgery subjects will have blood collected once at the start of surgery, once at the end of surgery, and once in the PACU. MRI patients will have blood collected once prior to the start of the MRI and once at the completion of the MRI.
Time Frame: On the day of surgery or MRI from start of procedure to discharge from PACU (approx. 1-7 hrs.)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MRI Control Arm
Number analyzed (Participants) | 25
pg/ml
  IL-1β pre-isoflurane | 25.97 (9.01)
  IL-1β post-isoflurane | 38.53 (16.56)
  TNF-α pre-isoflurane | 94.26 (18.07)
  TNF-α post-isoflurane | 85.84 (12.12)
  IL-6 pre-isoflurane | 2.28 (2.27)
  IL-6 post-isoflurane | 2.04 (2.15)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | MRI Control Arm
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT02512809/Prot_SAP_000.pdf